CLINICAL TRIAL: NCT05957094
Title: Human Cerebral Blood Flow and Serotonin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Phil Ainslie, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H23-01716
Record Dates: First submitted 2023-07-11; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Depression; Serotonin Deficiency
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Participants will complete all interventions (control and experimental) following drug washout
Who Masked: Participant, Investigator
Masking Description: The participant will not know whether they are receiving placebo or SSRI. The primary investigator will also no know if the participant is receiving placebo or SSRI
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo visit (Placebo Comparator): Participants will then undergo pre-intervention testing, with at least 20 minutes of rest between each. Once these tests are complete, the participant will ingest a placebo (sugar pill) that is identical in appearance to the drug condition. Three hours after placebo ingestion all tests will be conducted again. Participants will remain in the lab and will be free to read or work during this resting 3 hour period. This will conclude this experimental visit.
  Interventions: Other: Placebo
- SSRI visit (Active Comparator): Participants will then undergo pre-intervention testing, with at least 20 minutes of rest between each. Once these tests are complete, the participant will ingest citalopram (40 mg) Then three hours later all tests will be conducted again. Participants will remain in the lab and will be free to read or work during this resting 3 hour period. This will conclude this experimental visit.
  Interventions: Drug: Pharmacological agent: Citalopram

INTERVENTIONS:
Drug: Pharmacological agent: Citalopram — Participants will be given 40 mg in capsule form, which is a normal clinical dose.
  Arms: SSRI visit
Other: Placebo — Participants will ingest a placebo (sugar pill) that is identical in appearance to the drug condition.
  Arms: Placebo visit

SUMMARY:
Breathing, blood pressure, and blood flow into the brain are controlled - in part - by small areas in the brainstem; the central chemoreceptors. The mechanisms involved in the transmission of signals through the brainstem and also in controlling brain blood flow past the brainstem both use a molecule called serotonin. Citalopram is a "selective serotonin reuptake inhibitor" (or SSRI) which means it allows serotonin to be released in the brain but stops it from being reabsorbed. SSRIs are often used as antidepressants. This study aims to investigate the influence of an SSRI on the control of brain blood flow.

DETAILED DESCRIPTION:
PURPOSE To determine the influence of acute selective serotonin reuptake inhibition (SSRI) on cerebrovascular function in humans

HYPOTHESIS We hypothesize that SSRI will not impact CO2 reactivity (a measure of cerebral vascular function); will reduce neurovascular coupling (a measure of regional cerebral metabolism regulation of the vasculature), and will augment the ventilatory response to CO2 (a measure of brainstem chemosensitivity).

Justification:

There is ample evidence in animal models that the neurotransmitter serotonin (5-hydroxytryptamine; 5-HT) is an integral component in neuronal signalling in areas of the brainstem controlling ventilation, and that such 5-HT neurons directly innervate blood vessels and astrocytes (brain cells controlling blood flow) in the brainstem. Brainstem areas, in particular those of the raphe nuclei, containing 5-HT neurons, have been implicated as being actively involved with cerebral microvascular regulation. Extensive preclinical evidence suggests that 5-HT contributes directly to neurogenic control of the vascular beds surrounding raphe nuclei due to neuronal 5-HT release. Furthermore, increases in 5-HT can lead to an uncoupling of CBF and cerebral metabolism.

Increased 5-HT release or availability (e.g., through inhibition of reuptake) leads to a decrease in the relationship between CBF and cerebral metabolism, potentially indicating and impairment in the cerebral vasculature to respond to the needs of brain.

In humans, oral buspirone (a partial 5-HT agonist) decreases CBF in regions of the posterior cingulate while m-CPP (mixed 5-HT agonist/antagonist) increases the cerebral metabolic utilization of glucose (CMRglu) in several regions. Increases in CMRglu of 4% to 5% in the prefrontal cortex and relative decreases of 3% in occipitotemporal regions occur during oral fenfluramine (a 5-HT analogue; increases extracellular serotonin levels). Increases in CBF in the bilateral frontal cortex but decreases within the bilateral temporal cortex and left thalamus also occur in response to intravenous fenfluramine. Oral fenfluramine increases CMRglu in left prefrontal regions but CMRglu decreases in right hemispheric regions. Paroxetine - a commonly prescribed selective serotonin reuptake inhibitor (SSRI) - reduces resting cerebral perfusion especially in the brainstem. Finally, CMRglu is reduced in parts of the amygdala, hippocampus and striatum, and increases in the right superior parietal lobe, following oral fluoxetine. In summary, there is certainly modification of both CBF and CMRO2 with 5-HT perturbations, however, it is unclear whether cerebral vascular regulation per se is affected.

Intravenous infusion of ketanserin - a drug used to treat hypertension with its adrenergic receptor inhibition properties which also has some selective 5-HT2A receptor antagonist properties - is reported to have little effect on basal CBF, or cerebral defence against variations in partial pressure of arterial carbon dioxide (PaCO2) or blood pressure, but does reduce whole-brain cerebral O2 metabolism. However, ketanserin also elicits hypotension (lowered mean arterial pressure) that confounds analyses of CBF responses if not accounted for. Although serotonin per se has some vasoconstrictive effects, true SSRIs have little to no effects on blood pressure in humans, as such, it is difficult to assign these effects purely 5-HT related effects.

Serotonin is transported in circulation bound to platelets, and the release of this platelet-bound 5-HT is associated with increased immune responses (release of interleukin-6) from the vasculature. As such, there is precedent to assess the effects of SSRIs on platelet-bound and free plasma 5-HT, as well as adrenal cortisol secretion and immunological responses across the brain. This is relevant to the acute impacts of SSRIs on factors that contribute to lifetime cardiovascular health.

Almost 1 in 4 Canadians will suffer depression in the course of their lives. Although there has been recent dissention regarding the association between serotonin and depression , the prevalence of SSRIs is undeniable. Of North American adults diagnosed with depression, 61.6% use SSRIs; while between 2015 to 2018, ~13% of North Americans older than 18 reported taking antidepressant medications. Citalopram, a highly selective 5-HT reuptake inhibitor was has been prescribed to >30 million patients in >70 countries. Given the prevalence of SSRIs and the potential implications that 5-HT related neurovascular dysregulation may have for cerebral vascular function (and ventilation control and blood pressure control given the importance of 5-HT signalling in the brainstem) it is surprising that so little work has investigated the cerebral effects. There is little work in humans assessing the activity of serotonin in dynamic regulation of CBF. Cerebral responses to the five main drivers for which CBF is regulated [i.e., O2, CO2, mean arterial blood pressure, cerebral metabolism, and autonomic control], represent the functional reactivity of the cerebral vasculature. Measurement of these outcomes can give insight in to a number of vascular mechanisms and are widely used in research and clinical settings.

Although several studies have assessed basal steady state CBF and CMRO2 during 5-HT perturbations, none have investigated the effects of SSRI administration on cerebral vascular function as none have used CBF measurement techniques with sufficient temporal resolution to do so.

Research Design:

This study will be performed at the Centre for Heart, Lung and Vascular Health at the UBC Okanagan Campus. Participants will visit the laboratory on three occasions, the first of which should last ~30 minutes and rest of which should last no more than ~7 hours each; altogether totalling ~14.5 hours.

The first visit will consist of a familiarization visit wherein participants will be given all information regarding the study, and, should they give informed consent, will then have both ICAs and both VAs scanned using duplex ultrasound to assess patency of reliable images. Following the familiarisation, participants will visit the laboratory on two occasions, to undergo experimental visits which will include: a placebo visit and an SSRI visit. So that we can ensure full washout of SSRI between visits, the two experimental visits will be scheduled one week apart in males and one month apart in females (to account for menstrual cycle).

All participants will undergo all experimental sessions, in randomized, counterbalanced order. Participants will not be informed of which drug was received during which session until after the completion of the entire experimental study. Upon completion of informed written consent and the health questionnaire (submitted alongside this application) participants will be familiarized to the measurements and equipment.

STATISTICAL ANALYSES Differences in pre vs post test responses between visits will be examined using linear mixed modal analysis. Between-day variability of baseline responses will be examined using paired two-tailed T-tests. Repeatability between days within-subjects will be determined using Pearson's (r) and intraclass correlation coefficients (ICC2,1: two-way random effects, absolute agreement, single rater/measurement. Within-subjects coefficients of variation will be calculated for between-day assessments.

SAMPLE SIZE JUSTIFICATION There are no previous studies upon which to base a priori power calculations. As such, we estimate, based on previous studies from our laboratory assessing the same outcomes pre vs post other pharmacological interventions, that we will be adequately powered to see changes in cerebral variables from baseline with a sample size of n=~15.

ELIGIBILITY:
Inclusion Criteria:

* 15 healthy participants - mix of male and female - between 18 and 35 years of age will be recruited.

The maximum age of 35 was chosen so as to confine this study to "young adults", there is sufficient evidence to suggest that there is great variation of vascular responses to various stimuli across lifetime. As such, including participants from a larger range of ages would inevitably increase the physiological variability of the measures collected and thereby dilute the potential findings. Before assessing the effects of SSRI on CBF and ventilatory responses across the lifetime, we must first assess it in a single age-range cohort, to determine "young healthy normative" data.

Exclusion Criteria:

* Participants will be excluded from the study if they are:
* taking any medications,
* are or have recently (within the previous 6 months) been pregnant (self-reported - or pregnancy test result),
* currently smoke or smoked within the previous year,
* have had, or currently have cardiovascular, metabolic, respiratory, or neurological disease,
* are obese (BMI>30kg/m2),
* have had any invasive cerebral surgical procedures,
* have a cardiac pacemaker,
* we are unable to attain reliable ultrasound images of their neck arteries,
* currently or within the previous year have been prescribed SSRIs or other serotonergic drugs (tryptophan, triptans, lithium, fentanyl and its analogues, dextromethorphan, tramadol, tapentadol, meperidine, methadone and pentazocine or St. John's Wort),
* currently or within the previous year been prescribed monoamine oxidase inhibitors (another kind of anti-depressant),
* have recently (within the previous two weeks) used drugs including lysergic acid diethylamide (LSD), psilocybin (magic mushrooms), cocaine, or 3,4-Methylenedioxymethamphetamine (MDMA, ecstasy) (these drugs work via serotonin related mechanisms).

Both females and males will be tested. Contraceptive use will be noted but will not be part of any exclusion criteria. Phase of menstrual cycle will be noted but will not be part of any exclusion criteria, though females will be tested within the early follicular phase of menstruation, or the placebo phase of contraceptive use, and tested in the same (self-reported) phase of the next menstrual cycle.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Cerebral Blood Flow | Pre Citalopram
  Blood flow to the brain as measured using duplex ultrasonography
Cerebral Blood Flow | 3 hours following Citalopram
  Blood flow to the brain as measured using duplex ultrasonography
Exercise Performance | Pre Citalopram
  Maximum volume of oxygen consumed during maximal exercise
Exercise Performance | 3 hours following Citalopram
  Maximum volume of oxygen consumed during maximal exercise
Cerebrovascular reactivity to carbon dioxide | Pre Citalopram
  Cerebral blood flow response to increase in inspired carbon dioxide
Cerebrovascular reactivity to carbon dioxide | 3 hours following Citalopram
  Cerebral blood flow response to increase in inspired carbon dioxide

SECONDARY OUTCOMES:
Concentration of Platelet serotonin | Pre Citalopram
  Serotonin bound to platelets
Concentration of Platelet serotonin | 3 hours following Citalopram
  Serotonin bound to platelets

CONTACTS AND LOCATIONS:
Overall Officials: Philip Ainslie, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Okanagan Campus, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
No personal data will be made available publicly or to other researchers.